CLINICAL TRIAL: NCT05602675
Title: Evaluation of the Effect of LY3871801 on the Pharmacokinetics of CYP450 Substrates and an OAT1/3 Substrate in Healthy Participants
Brief Title: A Drug Interaction Study of LY3871801 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: 18336; J3P-MC-FTAD (Other: Eli Lilly and Company)
Record Dates: First submitted 2022-10-28; First posted 2022-11-02 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Healthy
MeSH Terms: interventions — Methotrexate; Warfarin; Dextromethorphan; Midazolam; repaglinide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LY3871801 + Methotrexate (Part 1) (Experimental): LY3871801 administered orally in combination with methotrexate given orally.
  Interventions: Drug: LY3871801; Drug: Methotrexate
- LY3871801 + Repaglinide + Drug Cocktail (Part 2) (Experimental): LY3871801 administered orally in combination with repaglinide given orally and drug cocktail which includes warfarin, dextromethorphan and midazolam administered orally.
  Interventions: Drug: LY3871801; Drug: Warfarin; Drug: Dextromethorphan; Drug: Midazolam; Drug: Repaglinide

INTERVENTIONS:
Drug: LY3871801 — Administered orally.
Drug: Methotrexate — Administered orally.
  Arms: LY3871801 + Methotrexate (Part 1)
Drug: Warfarin — Administered orally.
  Arms: LY3871801 + Repaglinide + Drug Cocktail (Part 2)
Drug: Dextromethorphan — Administered orally.
  Arms: LY3871801 + Repaglinide + Drug Cocktail (Part 2)
Drug: Midazolam — Administered orally.
  Arms: LY3871801 + Repaglinide + Drug Cocktail (Part 2)
Drug: Repaglinide — Administered orally.
  Arms: LY3871801 + Repaglinide + Drug Cocktail (Part 2)

SUMMARY:
The main purpose of this study is to determine the effect of LY3871801 when administered orally on the levels of methotrexate (part 1), drug cocktail (warfarin, dextromethorphan, and midazolam) and repaglinide (part 2) in the blood stream when administered orally in healthy participants. The information about any adverse effects experienced will be collected and the tolerability of LY3871801 will also be evaluated. The study may last up to approximately 25 days for each participant.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are overtly healthy as determined by medical evaluation including medical history and physical examination.
* Have body weight ≥ 45 kilograms (kg) and body mass index (BMI) within the range 18.5 to 40.0 kilograms per meter squared (kg/m²)
* Male or female participants not of childbearing potential (both parts) and for part 2, female participants of child bearing potential are eligible.

Exclusion Criteria:

* Have known allergies to LY3871801, related compounds, or any components of the formulation, or history of significant atopy.
* Have known allergies to drugs including methotrexate, folic acid, repaglinide, warfarin, dextromethorphan, and midazolam that would pose an unacceptable risk to the participant.
* Have an abnormal blood pressure and/or pulse rate, deemed to be clinically significant by the investigator
* Have used or intend to use prescription or nonprescription medication
* Have a positive (not indeterminate) QuantiFERON®-TB Gold test

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2022-11-02 (Actual); Primary Completion 2023-03-29 (Actual); Study Completion 2023-03-29 (Actual)

PRIMARY OUTCOMES:
Part 1: Pharmacokinetics (PK): Maximum Concentration (Cmax) of Methotrexate | Predose up to 48 hours postdose
  Part 1: PK: Cmax of Methotrexate
Part 1: PK: Area Under the Plasma Concentration Versus Time Curve From Zero to Infinity (AUC[0-∞]) of Methotrexate | Predose up to 48 hours postdose
  Part 1: PK: AUC[0-∞] of Methotrexate
Part 2: PK: Cmax of Midazolam | Predose up to 24 hours postdose
  Part 2: PK: Cmax of Midazolam
Part 2: PK: AUC[0-∞] of Midazolam | Predose up to 24 hours postdose
  Part 2: PK: AUC[0-∞] of Midazolam
Part 2: PK: Cmax of S-warfarin | Predose up to 96 hours postdose
  Part 2: PK: Cmax of S-warfarin
Part 2: PK: AUC[0-∞] of S-warfarin | Predose up to 96 hours postdose
  Part 2: PK: AUC[0-∞] of S-warfarin
Part 2: PK: Cmax of Dextromethorphan | Predose up to 72 hours postdose
  Part 2: PK: Cmax of Dextromethorphan
Part 2: PK: AUC[0-∞] of Dextromethorphan | Predose up to 72 hours postdose
  Part 2: PK: AUC[0-∞] of Dextromethorphan
Part 2: PK: Cmax of Repaglinide | Predose up to 24 hours postdose
  Part 2: PK: Cmax of Repaglinide
Part 2: PK: AUC[0-∞] of Repaglinide | Predose up to 24 hours postdose
  Part 2: PK: AUC[0-∞] of Repaglinide

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Covance Dallas, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No